CLINICAL TRIAL: NCT05935137
Title: Evaluation of Coagulation Status of Pregnant Women in the Peripartum Period Using the Device Clotpro®, a Prospective Observational Study
Brief Title: Evaluation of Coagulation Status of Pregnant Women in the Peripartum Period Using the Device Clotpro®
Status: Completed | Type: Observational
Sponsor: Ondrej Hrdy (Other)
Responsible Party: Sponsor-Investigator, Ondrej Hrdy, vice chair for education, Brno University Hospital
Organization: Brno University Hospital (Other)
Other Study IDs: 01-120423/EK
Record Dates: First submitted 2023-05-25; First posted 2023-07-07 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Coagulation and Hemorrhagic Disorders
Keywords: Blood coagulation; Fibrinogen; Viscoelastic method; Pregnancy; Labor
MeSH Terms: conditions — Thrombosis; Hemorrhagic Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pregnant women: It is a group of pregnant women after finished 37th week of gestation. We will take blood sample for a coagulation test on the device ClotPro.There is no more intervention.
  Interventions: Diagnostic Test: Coagulation test on device ClotPro
- Non-pregnant women: It is a control group - non-pregnant women. We will take blood samples for blood count and coagulation status and a coagulation test on the device ClotPro.There is no more intervention.
  Interventions: Diagnostic Test: Coagulation test on device ClotPro

INTERVENTIONS:
Diagnostic Test: Coagulation test on device ClotPro — The blood sample for coagulation test on device ClotPro will be take for both group and the test will be provided.

SUMMARY:
The primary aim of the study is to determine the physiological parameters of the coagulation status of pregnant women in the peripartum period (PWPP) for the ClotPro® device - Ex-test (CT, CFT, MCF, A5, A10, A20, ML), In-test (CT, CFT, MCF, A5, A10, A20, ML) and Fib-test (CT, CFT, MCF, A5, A10, A20, ML) and based on these results, establish ClotPro® reference ranges in parturients. The secondary aim is to compare the difference in coagulation parameters between pregnant women in the peripartum period and a control group of non-pregnant women (NPW) on the ClotPro® device. Furthermore, a comparison with the physiological parameters of pregnant women in the peripartum period intended for ROTEM® and TEG® devices (they are already known).

DETAILED DESCRIPTION:
This is a prospective observational cross-sectional study with a control group whose task is to describe the physiological parameters of the coagulation status of pregnant women in the peripartum period measured on the ClotPro® device. The study is monocentric and will take place at the Brno University Hospital. The study will evaluate a group of pregnant women in the peripartum period who come to give birth at the Brno University Hospital and fulfill the inclusion criteria, the target number is 120 patients. A control group of non-pregnant patients who fulfill the inclusion criteria to verify the difference between pregnant patients in the peripartum period and non-pregnant patients will also be included, the target number is 40 patients. For the participant the study is completed after obtaining the results from the ClotPro® device, there will be no reaction to result. The study is an academic research project, not sponsored by a private entity, and data will not be provided to a private entity.

The primary aim of the study is to determine the physiological parameters of the coagulation status of pregnant women in the peripartum period (PWPP) for the ClotPro® device - Ex-test (CT, CFT, MCF, A5, A10, A20, ML), In-test (CT, CFT, MCF, A5, A10, A20, ML) and Fib-test (CT, CFT, MCF, A5, A10, A20, ML) and based on these results, establish ClotPro® reference ranges in parturients. The secondary aim is to compare the difference in coagulation parameters between pregnant women in the peripartum period and a control group of non-pregnant women (NPW) on the ClotPro® device. Furthermore, a comparison with the physiological parameters of pregnant women in the peripartum period intended for ROTEM® and TEG® devices (they are already known).

ELIGIBILITY:
GROUP: Pregnant woman

Inclusion Criteria:

* Age 18 - 45 years
* BMI 18.5 - 30.0
* Negative pregnancy test
* The patient is able to sign an informed consent

Exclusion Criteria:

* Antiplatelet treatment
* Anticoagulation treatment
* Hereditary or acquired coagulopathy
* History of thrombosis or pulmonary embolism
* Acute or chronic inflammation (fever, septic condition, autoimmune disease)
* Active bleeding
* History of hemato-oncological disease
* Refusal of inclusion in the study by the patient

GROUP: Non-pregnant group

Inclusion Criteria:

* A pregnant woman admitted to Department of gynecology and obstetrics for the labor at the physiological term (38th week (38+0) and more)
* Age 18 - 45 years
* BMI 18.5 - 30.0 (before pregnancy)
* Blood samples are indicated for standard blood samples before labor
* The patient is able to sign an informed consent at the time of admission

Exclusion Criteria:

* Antiplatelet treatment
* Anticoagulation treatment
* Hereditary or acquired coagulopathy
* History of thrombosis or pulmonary embolism
* Acute or chronic inflammation (fever, septic condition, autoimmune disease)
* Active bleeding
* Preeclampsia
* Eclampsia
* Gestational diabetes
* Abruption of the placenta
* HELLP syndrome
* History of hemato-oncological disease
* Pregnancy in last 6 months
* Refusal of inclusion in the study by the patient

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: GROUP: Pregnant woman Population of pregnant women fulfilling all inclusion criteria and none of exclusion criteria.
  GROUP: Non-pregnant group Population of non-pregnant women fulfilling all inclusion criteria and none of exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

PRIMARY OUTCOMES:
CT for Ex-test on ClotPro® device | before the labor
  Clotting time for Ex-test ClotPro® device
CT for In-test on ClotPro® device | before the labor
  Clotting time for In-test ClotPro® device
CT for Fib-test on ClotPro® device | before the labor
  Clotting time for Fib-test ClotPro® device
CFT for Ex-test on ClotPro® device | before the labor
  Clot formation time for Ex-test ClotPro® device
CFT for In-test on ClotPro® device | before the labor
  Clot formation time for In-test ClotPro® device
CFT for Fib-test on ClotPro® device | before the labor
  Clot formation time for Fib-test ClotPro® device
A5 for Ex-test on ClotPro® device | before the labor
  Maximum clot firmness in 5th minute for Ex-test ClotPro® device
A5 for In-test on ClotPro® device | before the labor
  Maximum clot firmness in 5th minute for In-test ClotPro® device
A5 for Fib-test on ClotPro® device | before the labor
  Maximum clot firmness in 5th minute for Fib-test ClotPro® device
A10 for Ex-test on ClotPro® device | before the labor
  Maximum clot firmness in 10th minute for Ex-test ClotPro® device
A10 for In-test on ClotPro® device | before the labor
  Maximum clot firmness in 10th minute for In-test ClotPro® device
A10 for Fib-test on ClotPro® device | before the labor
  Maximum clot firmness in 10th minute for Fib-test ClotPro® device
A20 for Ex-test on ClotPro® device | before the labor
  Maximum clot firmness in 20th minute for Ex-test ClotPro® device
A20 for In-test on ClotPro® device | before the labor
  Maximum clot firmness in 20th minute for In-test ClotPro® device
A20 for Fib-test on ClotPro® device | before the labor
  Maximum clot firmness in 20th minute for Fib-test ClotPro® device
MCF for Ex-test on ClotPro® device | before the labor
  Maximum clot firmness for Ex-test ClotPro® device
MCF for In-test on ClotPro® device | before the labor
  Maximum clot firmness for In-test ClotPro® device
MCF for Fib-test on ClotPro® device | before the labor
  Maximum clot firmness for Fib-test ClotPro® device
ML for Ex-test on ClotPro® device | before the labor
  Maximum lysis for Ex-test ClotPro® device
ML for In-test on ClotPro® device | before the labor
  Maximum lysis for In-test ClotPro® device
ML for Fib-test on ClotPro® device | before the labor
  Maximum lysis for Fib-test ClotPro® device
Hemoglobin level | before the labor
  Hemoglobin level
Hematocrite level | before the labor
  Hematocrite level
Platelet level | before the labor
  Platelet level
Leucocytes level | before the labor
  Leucocytes level
Fibrinogen level | before the labor
  Fibrinogen level
Prothrombin time | before the labor
  Prothrombin time
activated Partial thromboplastin time | before the labor
  activated Partial thromboplastin time
INR | before the labor
  INR
Thrombin time | before the labor
  Thrombin time
Establish ClotPro® reference ranges in parturients | before the labor
  Reference ranges will be established according to IFCC guidelines, based on physiological coagulation parameters measured in parturient women using the ClotPro® device.

SECONDARY OUTCOMES:
Age | before the labor
  Age
Weight | before the labor
  Weight
Weight | before pregnancy
  Weight
Height | before the labor
  Height
BMI | before the labor
  BMI
BMI | before pregnancy
  BMI
Number of pregnancies | before the labor
  Number of pregnancies
Multiplicity of pregnancy | before the labor
  Multiplicity of pregnancy
Smoking | before the labor
  Smoking
Blood loss | immediately after the labor
  Blood loss
Type of labour | immediately after the labor
  spontaneous labor or cesarian section
Term of delivery | immediately after the labor
  Term of delivery
Comparison of fibrinogen level and Fib-test | before the labor
  Comparison of fibrinogen level and Fib-test
Comparison of Prothrombin time and CT in Ex-test | before the labor
  Camparison of Prothrombin time and CT in Ex-test
Comparison of activated Partial thromboplastin time and In-test | before the labor
  Comparison of activated Partial thromboplastin time and In-test

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gal, prof, Study Director — University Hospital Brno
Locations (1):
- University Hospital Brno, Brno, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Say L, Chou D, Gemmill A, Tuncalp O, Moller AB, Daniels J, Gulmezoglu AM, Temmerman M, Alkema L. Global causes of maternal death: a WHO systematic analysis. Lancet Glob Health. 2014 Jun;2(6):e323-33. doi: 10.1016/S2214-109X(14)70227-X. Epub 2014 May 5. PMID 25103301
- [Background] Ohno N, Fukamiya N, Okano M, Tagahara K, Lee KH. Synthesis of cytotoxic fluorinated quassinoids. Bioorg Med Chem. 1997 Aug;5(8):1489-95. doi: 10.1016/s0968-0896(97)00095-3. PMID 9313855
- [Background] Kietaibl S, Ahmed A, Afshari A, Albaladejo P, Aldecoa C, Barauskas G, De Robertis E, Faraoni D, Filipescu DC, Fries D, Godier A, Haas T, Jacob M, Lance MD, Llau JV, Meier J, Molnar Z, Mora L, Rahe-Meyer N, Samama CM, Scarlatescu E, Schlimp C, Wikkelso AJ, Zacharowski K. Management of severe peri-operative bleeding: Guidelines from the European Society of Anaesthesiology and Intensive Care: Second update 2022. Eur J Anaesthesiol. 2023 Apr 1;40(4):226-304. doi: 10.1097/EJA.0000000000001803. PMID 36855941
- [Background] Quinlan SM, Scalapino DJ. Neutron scattering from a dx2-y2-wave superconductor with strong impurity scattering and Coulomb correlations. Phys Rev B Condens Matter. 1995 Jan 1;51(1):497-504. doi: 10.1103/physrevb.51.497. No abstract available. PMID 9977110
- [Background] de Lange NM, van Rheenen-Flach LE, Lance MD, Mooyman L, Woiski M, van Pampus EC, Porath M, Bolte AC, Smits L, Henskens YM, Scheepers HC. Peri-partum reference ranges for ROTEM(R) thromboelastometry. Br J Anaesth. 2014 May;112(5):852-9. doi: 10.1093/bja/aet480. Epub 2014 Jan 31. PMID 24486836